CLINICAL TRIAL: NCT03406338
Title: Surgical Fasciectomy Versus Collagenase Injection in Treating Recurrent Dupuytren Disease: a Randomized Controlled Trial
Brief Title: Fasciectomy vs Collagenase Injection in Recurrent Dupuytren Disease
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Isam Atroshi, Professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hlm_DC
Record Dates: First submitted 2018-01-14; First posted 2018-01-23 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Dupuytren Disease of Finger
MeSH Terms: interventions — Fasciotomy; Surgical Procedures, Operative; Microbial Collagenase

STUDY DESIGN:
Intervention Model Description: Randomized parallel Group, ratio 1:1.
Who Masked: Outcomes Assessor
Masking Description: Before examination the patients will wear thin gloves in the treated hands to conceal possible surgical scars so the examiner will be blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Surgical fasciectomy (Active Comparator): Fasciectomy according to usual care (surgery), implying excision of Dupuytren's cords and tissues to release the finger joint contractures
  Interventions: Procedure: Fasciectomy
- Collagenase Clostridium Histolyticum (Experimental): Injection of 0.8 mg collagenase clostridium histolyticum into multiple spots in the Dupuytren cords followed by finger manipulation 1-2 days later to release the finger joint contractures
  Interventions: Drug: Collagenase Clostridium Histolyticum

INTERVENTIONS:
Procedure: Fasciectomy — Surgical excision of Dupuytren cords causing finger joint contractures. Surgery done under regional or general anesthesia. Additional procedures (such as capsulotomy or skin graft) done if surgeon deemed necessary.
  Other Names: Surgery
  Arms: Surgical fasciectomy
Drug: Collagenase Clostridium Histolyticum — Injection of Collagenase into the Dupuytren cord after local anesthesia (nerve block) followed 24-48 hours later by finger manipulation after local anesthesia
  Other Names: Non-surgical treatment
  Arms: Collagenase Clostridium Histolyticum

SUMMARY:
This randomized controlled trial will compare the outcome of surgery (fasciectomy) with that of local injection of Collagenase Clostridium Histolyticum in patients with recurrent finger joint contracture after previous treatment with Surgery, collagenase injection or needle fasciotomy. Half of the participants will be treated with surgery while the other half will receive collagenase injection.

DETAILED DESCRIPTION:
No definitive cure for Dupuytren disease (DD) currently exists and recurrence of finger contractures after treatment is common. Surgical fasciectomy is considered the standard treatment method for patients with recurrence. However, the procedure is associated with a high incidence of complications. Injection of Collagenase Clostridium Histolyticum into Dypuytren cords causing the contracture is a non-surgical treatment for DD and has been shown to be a safe and effective method. Most studies regarding collagenase injection have involved first-time treatment. Efficacy of collagenase injection in patients with recurrent DD, beyond the immediate effect, has not yet been determined. This randomized trial will compare the outcome of surgical fasciectomy and collagenase injection in treating patients with finger joints contracture due to recurrent DD. The study is a single-center randomized controlled trial. Patients referred to an orthopedic department are screened for eligibility. The inclusion criteria are recurrence of DD in one or more fingers after previous treatment with fasciectomy, collagenase injection or needle fasciotomy, a passive extension deficit ≥30 degrees in the metacarpophalangeal (MCP) and/or proximal interphalangeal (PIP) joint in a previously treated finger, and a palpable cord believed to cause the recurrent contracture. A total of 56 patients will be randomized (computer-generated randomization list, stratified according to type of previous treatment and affected finger), to either surgical fasciectomy or collagenase injection. A blinded hand therapist will measure range of motion (including active and passive extension deficit) at baseline and 3 months, 12 months, 24 months and 60 months after treatment. The primary outcomes are the total active extension deficit (MCP plus PIP) at 3 months and the proportion of patients with contracture worsening ≥20 degrees in the treated finger joint at 2 years compared to 3 months. The secondary outcomes include total passive extension deficit, the 11-item disabilities of the arm, shoulder and hand (QuickDASH) score, EuroQol 5-dimensions (EQ-5D) index, cold intolerance symptom severity score, palmar pain score, pain visual analog scale (VAS) score, satisfaction VAS score, adverse events and costs.

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment for recurrence of Dupuytren´s contracture in at least one finger.
* Passive extension deficit of 30 degrees or greater in the metacarpophalangeal and/or proximal interphalangeal joint in a finger previously treated with surgical fasciectomy, collagenase injections, or needle fasciotomy.
* Palpable cord in the palm and/or affected finger causing the recurrent contracture.
* No Surgery, collagenase injection or needle fasciotomy in the finger with recurrent contracture in the past 12 months.

Exclusion Criteria:

* Medical comorbidities that constitute a contraindication for surgical fasciectomy or collagenase injection.
* Signs of nerve or vascular injury in the affected finger.
* Osteoarthritis in the metacarpophalangeal and/or proximal interphalangeal joint joint in the affected finger
* Complications after the previous treatment, such as infection or complex regional pain syndrome (CRPS).
* Previous trauma or other surgery involving the affected finger.
* More than 2 previous surgeries, collagenase injections or needle fasciotomies in the affected finger.
* Examining surgeon deems further fasciectomy inappropriate or potentially associated with very high complication risk, for example in severe contracture and/or severe scarring after the previous surgeries and considers salvage procedures (such as amputation) as the more appropriate treatment.
* Patient refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Total active extension deficit (metacarpophalangeal plus proximal interphalangeal joints) | Change from baseline to 3 months
  Extension deficit of the metacarpophalangeal and interphalangeal joints of the treated finger measured with hand-held goniometer (0 degrees indicates no extension deficit)
Proportion of patients with worsening in total active extension deficit ≥20 degrees | 24 months compared to 3 months
  Extension deficit of the metacarpophalangeal and interphalangeal joints of the treated finger measured with hand-held goniometer (0 degrees indicates no extension deficit)

SECONDARY OUTCOMES:
11-item disabilities of the arm, shoulder and hand (QuickDASH) score | Change over time from from baseline, 3 weeks, 6 weeks, 3 months, 12 months, 24 months and 60 months
  A patient-reported outcome measure of activity limitations related to upper extremity disorders, with total score range from 0 (best) to 100 (worst)
EuroQoL 5-dimensions (EQ-5D) Index | Change over time from from baseline, 3 weeks, 6 weeks, 3 months, 12 months, 24 months and 60 months
  Health-status and quality-of-life patient-reported measure, consists of 5 items, a single weighted score, the EQ-5D index, is calculated from the 5 dimensions, ranging from -0.594 (worst) to 1.0 (perfect health)
Pain score | Change over time from from baseline, 3 weeks, 6 weeks, 3 months, 12 months, 24 months and 60 months
  Visual analog scale of pain in the treated hand, score range from 0 (best) to 100 (worst)
Satisfaction score | 3 weeks, 6 weeks, 3 months, 12 months, 24 months and 60 months
  Visual analog scale of patient satisfaction with treatment outcome, score range from 0 (best) to 100 (worst)
Adverse events | Anytime during 24 months after treatment
  All observed and reported adverse events will be recorded on a standard form. Serious adverse events include nerve, artery or tendon damage, deep infection, complex regional pain syndrome and any complications requiring surgery or hospital admission.
Costs | From baseline through 24 months
  Total treatment cost, direct (medications, surgery, materials, visits etc) and indirect (sick leave related to the treatment)
Total active motion | Change from baseline to 3 months, 12 months, 24 months and 60 months
  Sum of active range of motion of metacarpophalangeal, proximal intephalangeal and distal interphalangeal joints of the treated finger
Total active extension deficit (metacarpophalangeal plus proximal interphalangeal joints) | Change from baseline to 12 months, 24 months and 60 months
  Active extension deficit of the metacarpophalangeal and interphalangeal joints of the treated finger measured with hand-held goniometer (0 degrees indicates no extension deficit)
Proportion of patients with worsening in total active extension deficit ≥20 degrees | 60 months compared to 3 months
  Extension deficit of the metacarpophalangeal and interphalangeal joints of the treated finger measured with hand-held goniometer (0 degrees indicates no extension deficit)
Palmar pain score | Change over time from baseline to 3 weeks, 6 weeks, 3 months, 12 months, 24 months and 60 months.
  2-item scale inquiring about pain in the palm and related activity limitations, total score range 0 (best) to 100 (worst)
Cold intolerance symptom severity score | Change from baseline to 3 weeks, 6 weeks, 3 months, 12 months, 24 months and 60 months.
  6-item scale inquiring about symptoms of cold intolerance, total score range 4 (best) to 100 (worst)
Total passive extension deficit (metacarpophalangeal plus proximal interphalangeal joints) | Change from baseline to 24 months and 60 months
  Passive extension deficit of the metacarpophalangeal and interphalangeal joints of the treated finger measured with hand-held goniometer (0 degrees indicates no extension deficit)

CONTACTS AND LOCATIONS:
Overall Officials: Isam Atroshi, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Department of Orthopedics Hässleholm-Kristianstad, Hässleholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nordenskjold J, Lauritzson A, Walden M, Kopylov P, Atroshi I. Surgical fasciectomy versus collagenase injection in treating recurrent Dupuytren disease: study protocol of a randomised controlled trial. BMJ Open. 2019 Feb 25;9(2):e024424. doi: 10.1136/bmjopen-2018-024424. PMID 30808670